CLINICAL TRIAL: NCT04907240
Title: Observational GORE® VIABAHN® Endoprosthesis With PROPATEN Bioactive Surface (VSX) Global Registry
Brief Title: Observational GORE® VIABAHN® Endoprosthesis With PROPATEN Bioactive Surface Global Registry
Status: Active, not recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: VSX 20-03
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Artery Disease; Popliteal Aneurysm; Hemodialysis Access; Visceral Artery Aneurysms; Trauma Injury
Keywords: Viabahn; EVAR; Propaten; Iliac; SFA; SFA ISR; AV access; VAA; PAA; Trauma; Injury
MeSH Terms: conditions — Peripheral Arterial Disease; Popliteal Artery Aneurysm; Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Iliac: Subjects with de novo or restenotic lesions in the iliac arteries treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
- Superficial Femoral Artery (SFA): Subjects with de novo or restenotic lesions in the SFA and proximal popliteal arteries treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
- Superficial Femoral Artery (SFA) In-Stent Restenosis (ISR): Subjects with in-stent restenosis lesions in the SFA and proximal popliteal arteries treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
- AV access: Subjects with stenosis or thrombotic occlusion at the venous anastomosis of synthetic arteriovenous (AV) access graft and in the venous outflow of dialysis access circuits, including the central veins treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
- Popliteal Artery Aneurysms: Subjects with popliteal artery aneurysms treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
- Trauma/Injury: Subjects with traumatic or iatrogenic vessel injuries in arteries that are located in the chest cavity, abdominal cavity, or pelvis (except for aorta, coronary, innominate, carotid, vertebral, and pulmonary arteries) treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
- Visceral Artery Aneurysms: Subjects with isolated visceral artery aneurysms treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)
- Others: Subjects treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX) but do not fit any of the cohorts listed above.
  Interventions: Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)

INTERVENTIONS:
Device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX) — Intent to treat with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX) in the treatment of Peripheral Artery Disease as part of routine clinical practice.

SUMMARY:
Collect real-world post-market clinical follow-up data on patients treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX)

DETAILED DESCRIPTION:
This is an Observational, prospective, single-arm, multicenter, post-market registry to collect real-world post-market clinical follow-up data on patients treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX) for one of the following indications: Iliac, Superficial Femoral Artery (SFA), Superficial Femoral Artery In-stent restenosis (SFA ISR), Hemodialysis access (AV access), Visceral artery aneurysms (VAA), Trauma/Injury, Popliteal Artery Aneurysms (PAA), or Other. Approximately 35 sites in Europe will participate and a minimum of 614 patients will be enrolled in this registry. All consecutive patients meeting protocol selection criteria, consented, with an intention to be treated with the GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface (VSX) will be included and followed through one year for Trauma/Injury and other; three years for VAA; five years for Iliac, SFA, SFA ISR and AV access and ten years for PAA per institutional standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Signed informed consent form
3. Suitable for endovascular treatment with VSX based on treating physician's best medical judgment
4. Willingness of the patient to adhere to institutional standard of care follow-up requirements

Exclusion Criteria:

1. Non-compliant lesions where full expansion of an angioplasty balloon catheter is not achievable during pre-dilatation, or where lesions cannot be dilated sufficiently to allow passage of the delivery system.
2. Use of the VSX Device in lesions involving a major side branch that may be covered by the endoprosthesis.
3. Lesion(s) cannot be treated with available VSX Device sizes per current Instructions for Use (IFU).
4. Lesion requires treatment with an altered endoprosthesis or delivery system. (Do not cut the endoprosthesis. The endoprosthesis should only be placed and deployed using the supplied catheter system).
5. Previous or concurrent enrollment into this registry (e.g., previous enrollment into another treatment cohort or patient requires enrollment into more than one cohort) (Note: Only the first VSX treatment will be enrolled if concurrent VSX procedures are performed that would require enrollment into more than one cohort).
6. Participation in concurrent research study or registry which may confound registry results, unless approved by Gore.
7. Known hypersensitivity to heparin or a previous incident of Heparin-Induced Thrombocytopenia (HIT) type II.
8. Unable to tolerate antiplatelet therapy.
9. Patient has a non-controllable allergy to contrast or the VSX Device components.
10. Pregnant or breast-feeding female at time of informed consent signature.
11. Life expectancy < 12 months due to comorbidities.
12. Patient has other medical conditions which, as determined by the investigator, may confound the data interpretation (e.g., sepsis, thrombophilic diseases, connective tissue disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients presenting with an indication for endovascular repair of one of the eight indications (iliac, SFA, SFA ISR, VAA, PAA, Trauma/Injury, AV access and others) are eligible for screening for participation in the registry. Only patients who meet all inclusion and no exclusion criteria, and who consent to participate will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 614 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from Device-Related Serious Adverse Events (SAE) | 12 month
  No adverse event that is deemed to be device-related and serious assessed by the investigator by cohort

SECONDARY OUTCOMES:
Freedom from Device-Related Serious Adverse Events (SAE) for patients treated specifically with PAHR09-13 | 36 months
  Equivalent device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface devices with catalogue numbers PAHR09-13.
  No adverse event that is deemed to be device-related and serious assessed by the investigator by cohort
Freedom from Target Lesion Revascularization (TLR) for patients treated specifically with PAHR09-13 | 36 months
  Equivalent device: GORE® VIABAHN® Endoprosthesis with PROPATEN Bioactive Surface devices with catalogue numbers PAHR09-13.
  No surgical or percutaneous revascularization procedure of the original treated lesion
Primary patency for subjects treated in iliac | 60 months
  Blood flow through the target lesion without the need for repeat surgical or endovascular procedures
Freedom from major amputation for subjects treated in iliac | 60 months
  No amputation above the level of the ankle of the treated index limb
Freedom from Target Lesion Revascularization (TLR) for subjects treated in SFA de novo / restenotic and SFA ISR | 60 months
  No surgical or percutaneous revascularization procedure of the original treated lesion
Freedom from major amputations for subjects treated in SFA de novo / restenotic and SFA ISR | 60 months
  No amputation above the level of the ankle of the treated index limb
Access secondary patency for subjects treated in Hemodialysis Access | 60 months
  Blood flow through the original treated lesion with the use of an additional or secondary surgical or endovascular procedures after occlusion occurs, with freedom from device related abandonment.
  Secondary access patency is maintained if the patient can still dialyze through the access but has abandoned it for some other reason such as a transplant
Freedom from death of any cause for subjects treated in Hemodialysis Access | 60 months
  Patient is free from death of any cause (is alive)
Primary Patency for subjects treated in PAA | 120 months
  Blood flow through the target lesion without the need for repeat surgical or endovascular procedures
Limb Salvage for subjects treated in PAA | 120 months
  Absence of an amputation above the level of the ankle of the index limb
Primary Patency for subjects treated in VAA | 36 months
  Blood flow through the target lesion without the need for repeat surgical or endovascular procedures
Device-related thrombosis for subjects treated in VAA | 36 months
  Stent thrombosis deemed to be device-related as assessed by the Investigator.
Treated Lesion Primary patency for subjects treated in Trauma-Injury | 12 months
  Blood flow through the target lesion without the need for repeat surgical or endovascular procedures
Device-related thrombosis for subjects treated in Trauma-Injury | 12 months
  Stent thrombosis deemed to be device-related as assessed by the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, PhD, Principal Investigator — Rijnstate Hospital, Arnhem, The Netherlands
Locations (26):
- iD3 Medical cvba, Sint-Agatha-Berchem, Belgium
- France (5):
  - Centre Hospitalier Unversitaire d'Angers, Angers
  - Centre Hospitalier Regional Universitaire de Brest, Brest
  - Hopital Edouard Herriot (HCL), Lyon
  - Hospital Paris Saint-Joseph, Paris
  - Clinique RHENA, Strasbourg
- Germany (5):
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Marien Krankenhaus, Hamburg
  - University of Heidelberg, Heidelberg
  - Krankenhaus Reinbek St. Adolf-Stift, Reinbek
  - University Hospital Tuebingen, Tübingen
- Papageorgiou Hospital, Pávlos, Greece
- Italy (5):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Fondazione Poliambulanza, Brescia
  - S.C. Chirurgia Vascolare dell'A.O.U. di Modena, Modena
  - Ospedale San Giovanni Molinette, Torino
  - Dipartimento di Scienze Chirurgiche e Morfologiche, Varese
- Netherlands (2):
  - Rijnstate, Arnhem
  - Medical Center Leeuwarden, Leeuwarden
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Alvaro Cunqueiro Hospital, Vigo
- Sweden (2):
  - Skane University Hospital, Malmo
  - Karolinska University Hospital, Solna
- United Kingdom (3):
  - Southmead Hospital, Bristol
  - Greater Glasgow Health Board, Glasgow
  - Queen Elizabeth Hospital, London

IPD SHARING:
Plan to Share IPD: No